CLINICAL TRIAL: NCT00872820
Title: Neural Mediators of Behavior Therapy for Anxiety
Brief Title: Examining Long-Term Effects and Neural Mediators of Behavioral Treatments for Social Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michelle Craske, PhD, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21MH081299 (NIH); R21MH081299 (NIH); DATR A3-NSS
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety; Social Anxiety Treatment; Cognitive Therapy; Mindfulness; Social Phobia; Social Phobia Treatment
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Participants will receive standard cognitive behavioral therapy.
  Interventions: Behavioral: Cognitive behavioral therapy
- 2 (Experimental): Participants will receive acceptance- and commitment-based behavioral therapy.
  Interventions: Behavioral: Acceptance- and commitment-based behavioral therapy
- 3 (No Intervention): Participants will be placed on a waitlist for 3 months before being offered treatment.

INTERVENTIONS:
Behavioral: Acceptance- and commitment-based behavioral therapy — 12 weekly treatment sessions conducted individually with a therapist; strategies for dealing with anxiety will include mindfulness and acceptance of negative feelings
  Arms: 2
Behavioral: Cognitive behavioral therapy — 12 weekly treatment sessions conducted individually with a therapist; methods for dealing with anxiety will include cognitive and breathing strategies
  Arms: 1

SUMMARY:
This study will compare the effects that two types of behavioral therapy have on brain function in people with social anxiety disorder.

DETAILED DESCRIPTION:
Social anxiety disorder (SAD) is characterized by intense and debilitating anxiety in common social situations. Cognitive behavioral therapy (CBT) is a talking treatment that aims to reduce immediate anxiety symptoms. However, some anxiety symptoms and comorbid disorders not directly addressed by CBT may only improve in the short term, while recurring in the long term. Behavioral therapy based on acceptance and mindfulness is thought to have longer lasting effects, because this approach emphasizes accepting anxiety instead of controlling anxiety. This study will compare standard CBT to acceptance and commitment therapy (ACT), which uses acceptance and mindfulness, to determine which is more effective on both a short- and long-term basis. Participants with SAD will undergo brain scans to determine how the two therapies affect brain functioning.

Participation in this study will last 12 months. Participants with SAD will be randomly assigned to receive CBT, ACT, or a waitlist condition. Both CBT and ACT treatments will include 12 weekly sessions that will deal with objects and situations that provoke anxiety. All sessions will be audio- and videotaped. The waitlist group will complete weekly self-monitoring forms to track anxiety and panic and will receive a phone call from a research coordinator every 2 weeks to make sure symptoms have not worsened. After 12 weeks, participants on the waitlist will be offered treatment.

All participants will attend study visits to undergo brain scanning at baseline, after 3 months, and after 12 months. Each study visit will involve MRI scanning (to evaluate brain structure), functional MRI (fMRI) scanning (to evaluate brain function), questionnaires about a participant's experience in the scanner, and collection of saliva samples before, during, and after scanning. While undergoing the fMRI scan, participants will be asked to remain at rest for a certain period of time, and then to perform tasks that will engage certain parts of the brain. Assessments for all participants will occur at baseline and after 3, 6, and 12 months. These assessments will include diagnostic evaluations by a therapist, self-report questionnaires, ongoing self-monitoring, physiological measurements, cognitive assessments, and behavioral observation.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for social anxiety disorder
* Right-handed
* If taking medications, stabilized on current dose for 3 months
* If undergoing psychotherapy, stabilized for 6 months
* Speaks English

Exclusion Criteria:

* Currently undergoing cognitive behavioral therapy
* History of psychiatric hospitalization in the last 5 years
* Presence of serious medical condition, such as respiratory, cardiovascular, pulmonary, neurological, or muscular-skeletal disease or pregnancy
* Active suicidal ideation
* Current severe depression
* History of bipolar disorder, psychosis, mental retardation, or brain damage
* History of substance abuse or dependence in the last 6 months
* Presence of irremovable metal objects in the body that are not fMRI-safe
* Suffers from claustrophobia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Brain activity, assessed using functional magnetic resonance imaging (fMRI) | Measured at baseline and after 3 and 12 months

SECONDARY OUTCOMES:
Social anxiety symptoms | Measured at baseline and after 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michelle G. Craske, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Psychology Department - Franz Hall, Los Angeles, California, United States

REFERENCES:
- [Derived] Niles AN, Burklund LJ, Arch JJ, Lieberman MD, Saxbe D, Craske MG. Cognitive mediators of treatment for social anxiety disorder: comparing acceptance and commitment therapy and cognitive-behavioral therapy. Behav Ther. 2014 Sep;45(5):664-77. doi: 10.1016/j.beth.2014.04.006. Epub 2014 May 5. PMID 25022777